CLINICAL TRIAL: NCT03363009
Title: Contribution of Connected Devices in the Follow-up of the Observance of a Prehabilitation Program
Acronym: Prehab-Connect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical issues
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016/32; 2016- A01086-45 (Other: ANSM)
Record Dates: First submitted 2017-11-23; First posted 2017-12-05 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Surgery
Keywords: prehabilitation; connected devices
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected device with close following (Experimental): Data from connected devices (arm wrist watch, connected monitor of blood pressure, connected thermometer and pulse oximeter) will be analyzed every day and used for coaching
  Interventions: Device: Optimized group
- Connected device with standard coaching (Other): Data from connected devices (arm wrist watch, connected monitor of blood pressure, connected thermometer and pulse oximeter) will be saved but not used for coaching
  Interventions: Device: Control group

INTERVENTIONS:
Device: Optimized group — The data provided by the connected devices is analyzed daily; the patient receives a phone call in case of no realization of the objectives.
  Arms: Connected device with close following
Device: Control group — Data will be recorded but not analyzed daily during the period of participation. The patient receives a phone call one time a week to answer possible questions and modify the prescription of physical activity if need.
  Arms: Connected device with standard coaching

SUMMARY:
Poor physical performance and poor nutritional status increase the risk of complications after major surgery. Prehabilitation is the process of enhancing the functional capacity before surgery.

A major problem is the adherence of the patients to the physical program. A controlled randomized study is therefore proposed to determine the impact of coaching on functional exercise capacity. All patients will wear connected devices to measure their physical activity. They will be randomized to either a group in which coaching will be adapted to the physical activity, or a control group in which coaching is performed without any information about physical activity

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Patients scheduled for a surgical procedure 4 weeks later (more or less 1 week) after initial assessment
* Patients having consented to participate
* Patients benefiting from a social security system.

Exclusion Criteria:

* Pregnant or lactating women
* Inability to perform physical assessment
* Dependant patients
* Inability to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 2 months
  6 minutes walk test
Functional capacity | 2 months
  Maximal oxygen consumption

SECONDARY OUTCOMES:
Critical events | 2 months
  Number of critical events detected using the connected devices
Postoperative complications | 2 months
  Number of complication during the 2 months following surgery according to Dindo and Clavien classification

CONTACTS AND LOCATIONS:
Overall Officials: Barizien Nicolas, MD, Principal Investigator — Hopital Foch; Marc Fischler, Study Chair — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France